CLINICAL TRIAL: NCT02264938
Title: Drusen Morphology Changes in Nonexudative Age-related Degeneration Using Spectral Domain Optical Coherence Tomography After Oral Antioxidants Supplementation: One-year Results.
Brief Title: Drusen Morphology Changes in Nonexudative Age-related Degeneration After Oral Antioxidants Supplementation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Germans Trias i Pujol Hospital (Other)
Responsible Party: Principal Investigator, Xavier Valldeperas, MD, PhD, FEBO, Germans Trias i Pujol Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: AC-11-112
Record Dates: First submitted 2014-10-09; First posted 2014-10-15 (Estimated); Last update posted 2014-10-15 (Estimated); Status verified 2014-10

CONDITIONS: Macular Degeneration
MeSH Terms: conditions — Macular Degeneration | interventions — Antioxidants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Observation (No Intervention): Patients with AREDS category 2 and 3 AMD are observed during 1 year
- Antioxidant (Active Comparator): Patients with AREDS category 2 and 3 AMD are enrolled to take daily oral supplementation with lutein (12mg) + zeaxanthin (2mg) + astaxanthin (8mg) + omega-3 fatty acids (docosahexaenoic acid [DHA] 540mg + eicosapentaenoic acid [EPA] 360mg) + vitamin C (40mg) + vitamin E (20mg) + zinc (16mg) + copper (2mg) during 1 year.
  Interventions: Dietary Supplement: Antioxidant

INTERVENTIONS:
Dietary Supplement: Antioxidant — Oral supplemmentation with antioxidants
  Arms: Antioxidant

SUMMARY:
Purpose: To determine drusen morphology (volume and area) changes in nonexudative age-related macular degeneration (AMD) after one year of oral supplementation with AREDS-like formulation.

DETAILED DESCRIPTION:
Methods: Patients with AREDS category 2 and 3 AMD were prospectively enrolled in this study, and were randomized to receive daily oral supplementation with lutein (12mg) + zeaxanthin (2mg) + astaxanthin (8mg) + omega-3 fatty acids (docosahexaenoic acid [DHA] 540mg + eicosapentaenoic acid [EPA] 360mg) + vitamin C (40mg) + vitamin E (20mg) + zinc (16mg) + copper (2mg), or observation during one year. ETDRS vision, biomicroscopy, intraocular pressure (IOP), color fundus photography and automatic measurement of drusen with Topcon 3D-OCT 2000 (Topcon, Tokyo, Japan) using the 6 x 6 mm 3D cube scan protocol, were performed in all patients, at baseline and 12 months after. Automated delineation of macular drusen was modified by the investigators when evident segmentation errors occurred.

ELIGIBILITY:
Inclusion Criteria:

* AREDS category 2 and 3 AMD

Exclusion Criteria:

* AREDS category 4 AMD
* other ophthalmological diseases
* currently on antioxidant supplementation

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Actual)
Dates: Start 2013-01; Primary Completion 2014-07 (Actual); Study Completion 2014-10 (Actual)

PRIMARY OUTCOMES:
Drusen volume change | 12 months

REFERENCES:
- [Derived] Evans JR, Lawrenson JG. Antioxidant vitamin and mineral supplements for slowing the progression of age-related macular degeneration. Cochrane Database Syst Rev. 2023 Sep 13;9(9):CD000254. doi: 10.1002/14651858.CD000254.pub5. PMID 37702300